CLINICAL TRIAL: NCT06900361
Title: Feasibility and Acceptability of Asthma Self-Management Delivered Through a Mobile Phone Application: A Pilot Study in Malawi
Brief Title: Use of Mobile Phone Application for Asthma Sele Management
Status: Completed | Type: Observational
Sponsor: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: P.09/20/3132; 5U24HL136791 (NIH)
Record Dates: First submitted 2025-03-26; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Asthma Self Management
Keywords: Asthma Self Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aimed to assess the feasibility and acceptability of self-management provided through a mobile application.

DETAILED DESCRIPTION:
The chronic nature of asthma management requires a long-term approach taking into account the variability of disease symptoms, triggers and exacerbations. Several current guidelines advocate for self-management as part of standard care. Low-income countries (LMICs) such as Malawi are experiencing an increase in the burden of disease which hinders delivery of self-management services. Mobile phone health applications (mHealth) has been reported as an effective and cost-effective tool in the monitoring and management of asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 10 years and over
2. Have a Physician diagnosis of asthma and be prescribed a salbutamol inhaler
3. Reside in Blantyre
4. Participants should be able to read and write either English or Chichewa with Minimum standard 5 eductaion

Exclusion Criteria:

1. Cognitively impaired
2. Presence of coormobities
3. Refues to consent
4. Presence of active lung disease other than athsma

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All asthma patients aged 10 years and over attending pediatric outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
GINA Symptom Control Assessment | one year
  Asthma Control Test (ATC) Score

CONTACTS AND LOCATIONS:
Locations (1):
- Kamuzu University of Malawi, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
The de-identified datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year

REFERENCES:
- [Background] Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention,2019. Available from www.ginasthma.org
- See also: 8. Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention,2019 — https://ginasthma.org/